CLINICAL TRIAL: NCT04666285
Title: A Survey of Southampton Women's Survey Women's and Offspring's Health and Wellbeing During the COVID-19 Pandemic and Lockdown.
Brief Title: Southampton Women's Survey COVID-19 Study
Acronym: SWS_COVID-19
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: 56780
Record Dates: First submitted 2020-10-15; First posted 2020-12-14 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Experience of pandemic — Experience of the pandemic will be studied through online questionnaire responses

SUMMARY:
The current COVID-19 pandemic has brought many challenges with implications for wellbeing and mental health. The Southampton Women's Survey provides the opportunity to understand influences on these important outcomes amongst women and their offspring in the context of an established longitudinal cohort study.

DETAILED DESCRIPTION:
Between 1998 and 2002 the Southampton Women's Survey (SWS) team interviewed 12,583 Southampton women aged 20 to 34 years. The baseline survey collected data on women's diets, lifestyles, body and blood measures, reproductive health, education, mental health and social circumstances. Of these participants, 3,158 women subsequently became pregnant within the study period and delivered a liveborn singleton infant. The survey has followed up the offspring and mothers with home visits at six months, one, two and three years. A sample of over 1,000 offspring was seen at 4 years of age, more than 2,000 offspring were seen at ages 6-7 years, and more than 1,000 at 8-9 years. Follow-up of offspring aged 11-13 years is being completed and at 17-19 years is being piloted.

The women are currently aged 37 to 57 years and the offspring are currently aged 12 to 21 years.

The COVID-19 pandemic has brought unique challenges across the population. The effects include those of the threat of the virus itself as well as the impact of the government-imposed lockdown on health and wellbeing. Research in many contexts will allow greater understanding of the repercussions of this unprecedented event. The Southampton Women's Survey provides an opportunity to understand the effects of the lockdown on a well-characterised cohort of women and their adolescent/young adult offspring. The longitudinal data available in the cohort will provide a unique opportunity to understand how circumstances earlier in life (including pre-pregnancy) influence people's health and wellbeing during the pandemic.

Objectives:

1. To collect individual level data relating to health and wellbeing during the COVID-19 pandemic amongst SWS women and their offspring.
2. To assess whether lockdown-specific pressures such as working from home, home schooling and lack of social contact are associated with health and wellbeing during the pandemic.
3. To use longitudinal data to understand how health and lifestyle in earlier life (including pre-pregnancy) are associated with health and wellbeing during the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Women with offspring born in the Southampton Women's Survey (original project)
* Offspring born in the Southampton Women's Survey (original project)

Exclusion Criteria:

* anyone who was not a part of the original project

Ages: 12 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Between 1998 and 2002 the Southampton Women's Survey team interviewed 12,583 Southampton women aged 20 to 34 years. Of these participants, 3,158 women subsequently became pregnant within the study period and delivered a liveborn singleton infant.
Sampling Method: Non-Probability Sample
Enrollment: 832 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Mental Health in women | 3 months
  General Health Questionnaire (GHQ-12) - higher score more severe condition

SECONDARY OUTCOMES:
Mental Health in offspring | 3 months
  Warwick Edinburgh Mental Wellbeing Scale (WEMWBS) - higher score describes better mental health

CONTACTS AND LOCATIONS:
Overall Officials: Keith Godfrey, BM, PhD,FRCP, Principal Investigator — Professor of Human Development and Health
Locations (1):
- MRC Lifecourse Epidemiology Unit, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided